

# Clinical Development

#### ACZ885/Canakinumab

#### CACZ885N2301E2

# An extension study of CACZ885N2301, multi-center, open label study of canakinumab in patients with Periodic Fever Syndromes (TRAPS, HIDS, or crFMF)

Statistical Analysis Plan (SAP)

Author: Statistician,

Document type: SAP Documentation

Document status: Final 2.0

Release date: 12-September-2016

Number of pages: 15

Property of Novartis
For business use only
May not be used, divulged, published or otherwise disclosed
without the consent of Novartis

Novartis For business use only Page 2 SAP CACZ885N2301E2

# **Document History – Changes compared to previous final version of SAP**

| Date | Time | Reason for | Outcome for update | Section and title |
|------|-------|------------|--------------------|-------------------|
| | point | update | | impacted |
| | | | | (Current) |

| Та | | f conter | nts | 2 |
|---|---|---|---|---|
| | | | iations | |
| 1 | | | | |
| - | 1.1 | | lesign | |
| | | 1.1.1 | Screening epoch (Epoch 1) | |
| | | 1.1.2 | Extension-treatment epoch (Epoch 2) | |
| | | 1.1.3 | Sample size calculation | |
| | | 1.1.4 | Primary analysis time point | |
| | | 1.1.5 | Interim analysis | |
| | 1.2 | Study o | objectives and endpoints | |
| 2 | Statis | Statistical methods | | |
| | 2.1 | | Data analysis general information | |
| | | 2.1.1 | General definitions | 8 |
| | 2.2 | Analys | is sets | 8 |
| | | 2.2.1 | Subgroup of interest | 8 |
| | 2.3 | Patient | disposition, demographics and other baseline characteristics | 8 |
| | | 2.3.1 | Patient disposition | 8 |
| | 2.4 | | nents (study treatment, rescue medication, concomitant therapies, ance) | g |
| | | 2.4.1 | Study treatment / compliance | |
| | | 2.4.2 | Prior, concomitant and post therapies | |
| | | | is of the primary objective | |
| | | 2.5.1 | Primary endpoint | 9 |
| | | 2.5.2 | Statistical hypothesis, model, and method of analysis | |
| | | 2.5.3 | Handling of missing values/censoring/discontinuations | |
| | | 2.5.4 | Supportive analyses | 9 |
| | 2.6 | Analys | is of the key secondary objective | 9 |
| | | 2.6.1 | Key secondary endpoint | 9 |
| | | 2.6.2 | Statistical hypothesis, model, and method of analysis | 9 |
| | | 2.6.3 | Handling of missing values/censoring/discontinuations | 10 |
| | 2.7 | Analysis of secondary efficacy objective(s) | | 10 |
| | | 2.7.1 | Secondary endpoints | 10 |
| | | 2.7.2 | Statistical hypothesis, model, and method of analysis | 10 |
| | | 2.7.3 | Handling of missing values/censoring/discontinuations | 10 |
| | 2.8 | Safety | analyses | 10 |
| | | 2.8.1 | Adverse events (AEs) | 10 |

| | | 2.8.2 | Deaths | 10 |
|---|-------|--------------------|----------------------------------------|----|
| | | 2.8.3 | Laboratory data | 10 |
| | | 2.8.4 | Other safety data | 10 |
| | 2.9 | Pharma | acokinetic endpoints | 11 |
| | 2.10 | PD and | PK/PD analyses | 11 |
| | 2.11 | Patient- | -reported outcomes | 11 |
| | 2.12 | Biomar | kers | 11 |
| | 2.13 | Other E | Exploratory analyses | 11 |
| | 2.14 | Interim | analysis | 11 |
| 3 | Samp | le size ca | llculation | 11 |
| 4 | Chang | ge to prot | tocol specified analyses | 11 |
| 5 | Appe | ndix | | 12 |
| | 5.1 | Imputa | tion rules | 12 |
| | | 5.1.1 | Study drug | 12 |
| | | 5.1.2 | AE date imputation | 12 |
| | | 5.1.3 | Concomitant medication date imputation | 12 |
| | 5.2 | AEs co | ding/grading | |
| | 5.3 | Labora | tory parameters derivations | 12 |
| | | 5.3.1 | Clinically notable laboratory values | |
| | 5.4 | Statistical models | | |
| | | 5.4.1 | Primary analysis | 15 |
| | | 5.4.2 | Key secondary analysis | |
| | 5.5 | Rule of | f exclusion criteria of analysis sets | |
| 6 | Refer | | | |
| | _ | | | |

Novartis For business use only Page 5 SAP CACZ885N2301E2

#### List of abbreviations

AE Adverse event

ALP Alkaline Phosphatase ALT Area Under the Curve

AST Aspartate Aminotransferase

crFMF colchicine resistant Familial Mediterranean Fever

CTC Common Toxicity Criteria

CTCAE Common Terminology Criteria for Adverse Events

ECG Electrocardiogram
HIDS Hyper IgD Syndrome

MedDRA Medical Dictionary for Drug Regulatory Affairs
PGA Physician's Global Assessment of Disease Activity

PSW Premature Subject Withdrawal

q4w Every 4 weeks q8w Every 8 weeks

SAE Serious Adverse Event

TBL Total Bilirubin

TD Study Treatment Discontinuation

TRAPS TNF-receptor Associated Periodic Syndrome

SAP Statistical Analysis Plan

#### 1 Introduction

This Statistical Analysis Plan (SAP) describes the plan for producing specific listings for study CACZ885N2301E2, which was planned to provide specific paients with opportunity to have access with canakinumab until approval in Japan.

The details about the study can be found in the latest version of the study protocol.

#### 1.1 Study design

Japanese patients are allowed to enter this extension study after completion of Epoch 4 (an open-label treatment epoch) in CACZ885N2301 study. This study consists of two study epochs (Screening epoch and Extension-treatment epoch). This study will be continued until approval of Canakinumab in Japan or the termination of the development of the Canakinumab in Periodic Fever Syndromes in Japan.

In this study, all patients will receive the same dose and regimen as administered at the end of study CACZ885N2301 consisting of 1 or 2 subcutaneous injections every 4 or 8 weeks. Safety will be evaluated every 8 weeks.

#### 1.1.1 Screening epoch (Epoch 1)

At Visit 1, patients will be assessed for eligibility for study participation after completion of Epoch 4 of the CACZ885N2301 study.

Visit 1 of this extension study and Visit 399 of the CACZ885N2301 study are conducted on the same day.

#### 1.1.2 Extension-treatment epoch (Epoch 2)

Patients who meet entry criteria at Visit 1 will enter the extension-treatment epoch (epoch 2). Since eligible patients initiate the extension- treatment epoch on the same day of screening, their first two visits (Visit 1 and Visit 101) can be on the same day.

Patients will continue the study drug based on the final dose and regimen administered at the end of the CACZ885N2301 study. All patients will receive 1 or 2 ACZ885 subcutaneous injections every 4 or 8 weeks. Stepwise up-titration up to a dosing regimen of ACZ885 300 mg (or 4 mg/kg for patients weighing  $\leq$  40 kg) every 4 weeks (q4w) will be allowed. In case of reflare [Physician's global assessment of disease activity (PGA)  $\geq$  2 AND CRP  $\geq$  30 mg/L], patients will be allowed to increase the dose as follows accordingly to the same up-titration scheme in study CACZ885N2301: If flare occurs at the last visit (V399) or visit between V309 and V399 of CACZ885N2301 study, up-titration will be allowed at visit 101.

- If patients receive ACZ885 150 mg (or 2 mg/kg for patients weighing  $\leq$  40 kg) every 8 weeks (q8w), they will increase the dose to ACZ885 150 mg q4w.
- If patients receive ACZ885 150 mg (or 2 mg/kg for patients weighing ≤ 40 kg) q4w, they will increase the dose to ACZ885 300 mg q4w.
- If patients receive ACZ885 300 mg (or 4 mg/kg for patients weighing ≤ 40 kg) q8w, they will increase the dose to ACZ885 300 mg q4w.

If flare occurs at the last visit (V399) it will be recorded in the CACZ885N2301 study. Safety will be evaluated every 8 weeks in the extension-treatment epoch (epoch 2). Patients receiving ACZ885 q4w or up-titrated to q4w administration, will come back every 4 weeks for unscheduled visits in addition to the scheduled visits.

For all patients, a safety follow-up visit should be conducted (e.g. by telephone) 30 days after study treatment discontinuation (TD)/ premature subject withdrawal (PSW), or 8 weeks after last injection of investigational drug, whichever is later.

#### 1.1.3 Sample size calculation

See section 3 "Sample size calculation".

#### 1.1.4 Primary analysis time point

No specific time point is considered as the one for primary analysis.

#### 1.1.5 Interim analysis

No interim analysis is planned.

#### 1.2 Study objectives and endpoints

The primary objective of this study is to evaluate safety and tolerability of ACZ885 in this extension study.

#### 2 Statistical methods

#### 2.1 Data analysis general information

All analyses for this study will be performed by Novartis using SAS version 9.4 or later.

For this study, only specific listings will be produced, and there will be no statistical summary presented.

All data will be presented for each individual cohorts, TRAPS, HIDS, and crFMF.

#### 2.1.1 General definitions

Table 2-1 General definitions

| Terms | Definiton |
|---|---|
| Study treatment | The treatment by dosing the investigational drug, canakinumab. |
| Date of first administration of extension treatment | The first visit date that the study treatment is given for this extension study. |
| Date of last administration of study treatment | The last visit date that the study treatment is given. |
| Extension Day 1 | Date of first administration of extension treatment |
| Extension Study Day | Extension Study Day is defined as (Event start date) – (Extension Day 1) + 1 for any event dated on or after Extension Day 1, or (Event start date) – (Extension Day 1) for any event dated before Extension Day 1. |
| Baseline | The last assessments obtained before the first dose of study treatment. This definition will be applied to percent change for creatinine clearance. |

#### 2.2 Analysis sets

The **Safety Set** will consist of all patients receiving at least one dose of study medication in the extension study.

#### 2.2.1 Subgroup of interest

Not applicable.

# 2.3 Patient disposition, demographics and other baseline characteristics

Patient demographic and baseline characteristic data to be collected on all patients include: date of birth, age, sex, race, ethnicity, relevant medical history/ current medical condition present before signing informed consent. Where possible, diagnoses but not symptoms will be recorded.

Demographic and baseline characteristics will be listed.

Any significant prior or active medical condition at the time of signing informed consent will be also listed.

#### 2.3.1 Patient disposition

The following listings will be presented:

- Subjects who discontinued prior to Epoch 2 on Safety Set
- Study completion during Epoch 2 on Safety Set

# 2.4 Treatments (study treatment, rescue medication, concomitant therapies, compliance)

#### 2.4.1 Study treatment / compliance

Exposure to study treatment will be listed. Also, the number of doses will be listed for individual patients.

For each patient, duration of exposure will be defined as (date of last visit in study) – (date of first administration of extension treatment) + 1.

#### 2.4.2 Prior, concomitant and post therapies

Listings will be provided to display prior/concomitant medications or therapies, and medical surgeries and procedures. Specifically, rescue medications will be listed.

Prior medications will be defined as treatments taken and stopped prior to date of first administration of study treatment. Any medication will be defined as a concomitant medication, if it is given at least once on or after date of first administration of study treatment.

Rescue medications will be defined as corticosteroids or NSAIDS provided as concomitant medications.

#### 2.5 Analysis of the primary objective

#### 2.5.1 Primary endpoint

The primary variable is adverse event. Details will be discussed in section 2.8.1.

#### 2.5.2 Statistical hypothesis, model, and method of analysis

Not applicable.

#### 2.5.3 Handling of missing values/censoring/discontinuations

Not applicable.

#### 2.5.4 Supportive analyses

Not applicable.

#### 2.6 Analysis of the key secondary objective

#### 2.6.1 Key secondary endpoint

Not applicable.

#### 2.6.2 Statistical hypothesis, model, and method of analysis

Not applicable.

#### 2.6.3 Handling of missing values/censoring/discontinuations

Not applicable.

#### 2.7 Analysis of secondary efficacy objective(s)

#### 2.7.1 Secondary endpoints

Not applicable.

#### 2.7.2 Statistical hypothesis, model, and method of analysis

Not applicable.

#### 2.7.3 Handling of missing values/censoring/discontinuations

Not applicable.

#### 2.8 Safety analyses

All safety analysis will be based on Safey Set.

#### 2.8.1 Adverse events (AEs)

A listing will be presented to display individual adverse events reported in Epoch 1 and 2.

Also, SAEs will be listed.

#### 2.8.1.1 Adverse events of special interest / grouping of AEs

Due to very much limited number of patients, no listing will be produced to display any grouping of AE.

#### 2.8.2 **Deaths**

Deaths will be listed.

#### 2.8.3 Laboratory data

All laboratory evaluations will be conducted locally.

Laboratory evaluations will be listed by patient. Additionally, notable abnormalities will be listed. Notable criteria will be defined as listed in section 5.3.1.

#### 2.8.4 Other safety data

#### 2.8.4.1 ECG and cardiac imaging data

Not applicable.

#### 2.8.4.2 Vital signs

Not applicable.

# 2.9 Pharmacokinetic endpoints

Not applicable.

## 2.10 PD and PK/PD analyses

Not applicable.

#### 2.11 Patient-reported outcomes

Not applicable.

#### 2.12 Biomarkers

Not applicable.

#### 2.13 Other Exploratory analyses

Not applicable.

#### 2.14 Interim analysis

No interim analysis is planned.

# 3 Sample size calculation

Patients who completed Epoch 4 of the preceding CACZ885N2301 study in Japan will be entered into this extension study. Therefore the maximum number of patients is 10.

# 4 Change to protocol specified analyses

Not applicable.

## 5 Appendix

#### 5.1 Imputation rules

Not applicable.

#### 5.1.1 Study drug

Not applicable.

#### 5.1.2 AE date imputation

Not applicable.

#### 5.1.3 Concomitant medication date imputation

Not applicable.

#### 5.1.3.1 Prior therapies date imputation

Not applicable.

#### 5.1.3.2 Post therapies date imputation

Not applicable.

#### 5.1.3.3 Other imputations

Not applicable.

#### 5.2 AEs coding/grading

Adverse events will be coded using MedDRA dictionary.

#### 5.3 Laboratory parameters derivations

#### 5.3.1 Clinically notable laboratory values

#### Notable laboratory abnormalities in adult patients (≥ 18 years of age)

Post-baseline values will be flagged as notable abnormalities as follows:

#### **Biochemistry**

- 1. ALT (SGPT): > 3 x, 5 x, 10 x, and 20 x Upper Limit of Normal (ULN) <sup>1</sup>
- 2. AST (SGOT):  $> 3 \text{ x}, 5 \text{ x}, 10 \text{ x}, \text{ and } 20 \text{ x ULN}^{-1}$
- 3. Elevation of AST and/ or ALT (> 3 x ULN) accompanied by elevated bilirubin (> 1.5 x ULN, > 2 x ULN)  $^{1}$
- 4. Any elevations of bilirubin; elevated total bilirubin (TBL) to  $> 2 \times ULN^{-1}$
- 5. Any elevations of ALP  $> 1.5 \times ULN^{-1}$
- 6. Gamma-Glutamyltransferase (GGT): > 3 x ULN

- 7. Creatinine (serum):  $\geq 3 \times ULN$
- 8. Creatinine clearance (CrCl) (Cockroft-Gault formula)  $^2$ :  $\geq 25\%$  decrease from baseline
- 9. Triglycerides: > 5 x ULN

#### Hematology

- 1. Hemoglobin:  $\geq 20$  g/L decrease from baseline or < 100 g/L
- 2. Platelet count<sup>3</sup>
  - CTC Grade 1: < Lower Limit of Normal (LLN) 75 x  $10^9$ /L
  - CTC Grade 2:  $< 75 50 \times 10^9/L$
  - CTC Grade 3:  $< 50 25 \times 10^9/L$
  - CTC Grade 4:  $< 25 \times 10^9/L$
- 3. White blood cell count <sup>3</sup>
  - CTC Grade 1: < LLN  $3 \times 10^9$ /L
  - CTC Grade 2:  $< 3 2 \times 10^9/L$
  - CTC Grade  $3: < 2 1 \times 10^9/L$
  - CTC Grade 4:  $< 1 \times 10^9/L$
- 4. Absolute neutrophils <sup>3</sup>
  - CTC Grade 1: < LLN  $1.5 \times 10^9$ /L
  - CTC Grade 2:  $< 1.5 1 \times 10^9/L$
  - CTC Grade 3:  $< 1 0.5 \times 10^9/L$
  - CTC Grade 4:  $< 0.5 \times 10E^9/L$
- 5. Absolute lymphocytes: < LLN
- 6. Absolute eosinophils:  $\geq 2.5 \text{ x}, \geq 3 \text{ x ULN}$

#### Urinalysis

Protein urine dipstick: ≥ ++

#### Notable laboratory abnormalities in pediatric patients (< 18 years of age)

Post-baseline values in pediatric patients (at the time of the assessment) will be flagged as notable abnormalities as follows:

#### **Biochemistry**

- 1. ALT (SGPT): > 3 x, 5 x, 10 x, and 20 x Upper Limit of Normal (ULN) <sup>1</sup>
- 2. AST (SGOT): > 3 x, 5 x, 10 x, and 20 x ULN <sup>1</sup>
- 3. Elevation of AST and/ or ALT (> 3 x ULN) accompanied by elevated bilirubin (> 1.5 x ULN, > 2 x ULN)  $^{1}$
- 4. Any elevations of bilirubin; elevated total bilirubin (TBL) to  $> 2 \times ULN^{-1}$
- 5. Any elevations of ALP  $> 1.5 \times ULN^{-1}$
- 6. GGT:  $\geq$  3 x, 5 x ULN
- 7. Creatinine (serum):  $\geq 1.5 \text{ x ULN}$
- 8. Creatinine clearance (Schwartz formula <sup>4</sup>): ≥ 25% decrease from baseline, ≥ 2 consecutive visits
- 9. Total Cholesterol: > 1.5 x ULN
- 10. Triglycerides:  $\geq 5.7 \text{ mmol/L}$
- 11. Creatinine clearance (Schwartz formula  $^4$ ):  $\geq 25\%$  decrease from baseline for  $\geq 3$  months in duration in combination with protein urine dipstick resulting in new protein  $\geq 1+, \geq 3$  months in duration

#### Hematology

- 1. Hemoglobin:  $\geq$  20 g/L decrease from baseline or < 85 g/L (patients < 16 years of age) or < 100 g/L (patients  $\geq$  16 years of age)
- 2. Platelet count<sup>3</sup>
  - CTC Grade 1: < Lower Limit of Normal (LLN) 75 x  $10^9$ /L
  - CTC Grade 2:  $< 75 50 \times 10^9/L$
  - CTC Grade 3:  $< 50 25 \times 10^9 / L$
  - CTC Grade 4:  $< 25 \times 10^9/L$
- 3. White blood cell count <sup>3</sup>
  - CTC Grade 1: < LLN 3 x  $10^9$ /L
  - CTC Grade 2:  $< 3 2 \times 10^9/L$
  - CTC Grade 3:  $< 2 1 \times 10^9/L$
  - CTC Grade 4:  $< 1 \times 10^9/L$
- 4. Absolute neutrophils <sup>3</sup>
  - CTC Grade 1: < LLN  $1.5 \times 10^9$ /L
  - CTC Grade 2:  $< 1.5 1 \times 10^9/L$
  - CTC Grade 3:  $< 1 0.5 \times 10^9/L$
  - CTC Grade 4:  $< 0.5 \times 10E^9/L$
- 5. Absolute lymphocytes: < LLN

6. Absolute Eosinophils:  $\geq 1.1 \text{ x ULN}$ ,  $\geq 0.45 \text{ x } 10^9/\text{L}$ 

#### Urinalysis

Protein urine dipstick:  $\geq$ + for  $\geq$  3 months in duration

#### 5.4 Statistical models

#### 5.4.1 Primary analysis

Not applicable.

#### 5.4.2 Key secondary analysis

Not applicable.

# 5.5 Rule of exclusion criteria of analysis sets

Table 5-1 Protocol deviations that cause subject to be excluded

| Deviation ID | Description of deviation | Exclusion from analysis |
|---|---|---|
| INCL02 | No written informed consent was obtained before any asessments were performed | Excluded from all analysis |
| TRT01 | Patient was not exposed to study medication at any visit | Excluded from analysis based on Safety Set |

#### 6 Reference

Schwartz GJ, Munoz A, Schneider MF, et al (2009) New Equations to Estimate GFR in Children with CKD. J Am Soc Nephrol; 20(3):629-37.

<sup>&</sup>lt;sup>1</sup> Adapted from FDA Guidance for Industry Drug-Induced Liver Injury: Premarketing Clinical Evaluation (July 2009)

<sup>&</sup>lt;sup>2</sup> Cockroft-Gault formula (Men): CrCl (mL/min) =  $[((140\text{-age (years})) \times \text{weight (kg)})/(\text{serum creatinine (}\mu\text{mol/L})/88.4) (\text{mg/dL}) \times 72]$ 

<sup>&</sup>lt;sup>2</sup> Cockroft-Gault formula (Women): CrCl (mL/min) =  $[((140\text{-age (years})) \times \text{weight (kg)})/(\text{serum creatinine }(\mu\text{mol/L})/88.4) (\text{mg/dL}) \times 72] \times 0.85$ 

<sup>&</sup>lt;sup>3</sup> Common Terminology Criteria for Adverse Events, US Department of Health and Human Services (v4.03: 14-Jun-2010)

<sup>&</sup>lt;sup>4</sup> Creatinine clearance was derived using the following formula: CrCl(mL/min/1.73 m2) = [0.413 x length (cm)/(serum creatinine mg/dl)] (Schwartz et al 2009)